CLINICAL TRIAL: NCT03600363
Title: A Prospective Randomized Controlled Phase II Clinical Trial of Metformin in the Maintenance Therapy of High Risk Diffuse Large B Lymphoma / Stage III Follicular Lymphoma Patients With Complete Remission
Brief Title: A Clinical Trial of Metformin in the Maintenance of Non-Hodgkin's Lymphoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Deputy Director of Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ-NHL-1805
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Stage III Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin arm (Experimental)
  Interventions: Drug: Metformin
- control arm (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Metformin — metformin (1.0g, bid) as a maintenance therapy in patients with complete remission
  Arms: metformin arm
Drug: Placebos — oral placebos as a maintenance therapy
  Arms: control arm

SUMMARY:
The study is to evaluate the therapeutic effect of metformin as a maintenance therapy in high risk patients with complete remission of diffuse large B lymphoma / stage III follicular lymphoma after chemotherapy in the initial R-CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone, plus the monoclonal antibody rituximab) regimen

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient age >14 years old;
2. Pathological types include: diffuse large B lymphoma, and stage III follicular lymphoma;
3. At the initial stage of therapy, received standard R-CHOP regimen and complete remission after the first course of treatment;
4. After complete remission, not consider to receive hematopoietic stem cell transplantation or chimeric antigen receptor T cell immunotherapy;
5. Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) not exceed 2 times of the normal upper limit;
6. Serum total bilirubin and creatinine not exceed 1.5 times of the normal upper limit;
7. Serum creatinine not exceed 1.5mg/dl;
8. Patients with high risk factors, including age > 60 year, or with diabetes/ impaired glucose tolerance, or with International Prognostic Index (IPI) score ≥2.
9. Sign informed consent file.

Exclusion Criteria:

1. Past medical history of high doses of cytarabine, methotrexate and rituximab maintenance therapy;
2. Past medical history of any type of hematopoietic stem cell transplantation;
3. Past medical history of lactic acidosis;
4. Extreme weight loss failure, malnutrition or dehydration patients;
5. Pregnant women or lactating women, or women who do not take contraceptive measures for childbearing age;
6. Alopecia, mental retardation or psychiatric disorders that affect the patient's normal informed consent;
7. Type 1.2 diabetes with ketoacidosis, liver function or renal insufficiency, pulmonary insufficiency, heart failure, acute myocardial infarction, severe infection and trauma, major surgery and clinical hypotension or hypoxia;
8. Diabetes complicated with severe chronic complications (such as diabetic nephropathy, diabetic retinopathy);
9. Any other serious complications occurred, depending on the outcome of the study;
10. Before the intravenous pyelography or anterior angiography;
11. Alcoholics;
12. Deficiency of Vitamin B12, folic acid or iron.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization until the date of trail closed or date of death from any cause, whichever came first, up to 100 months

SECONDARY OUTCOMES:
Progress Free Survival | From date of randomization until the date of trail closed or disease progressed, whichever came first, up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China